CLINICAL TRIAL: NCT05184387
Title: A Prospective Epidemiological Cohort Study Evaluating Occurrences of Influenza-like Illness in an Urban and Suburban Population of Healthy Subjects Aged 18-55 Years, Not Vaccinated Against Influenza.
Brief Title: A Prospective Epidemiological Cohort Study Evaluating Occurrences of Influenza-like Illness.
Status: Completed | Type: Observational
Sponsor: Osivax (Industry)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: OVX-FLU-001
Record Dates: First submitted 2021-11-26; First posted 2022-01-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples (total volume approximately 10 mL of whole blood per visit) obtained at study entry (before onset of the influenza season) and 6 months after, upon completion of the influenza season, will serve as alternative method for case confirmation and detection of unrecognized or asymptomatic infections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective epidemiological cohort: Urban and suburban population of healthy subjects aged 18-55 years, not vaccinated against influenza
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Collection of blood samples and completion of an electronic Diary (eDiary)

SUMMARY:
This Prospective epidemiological cohort study is being conducted in order to generate epidemiological data in support of Osivax's clinical development of a broad spectrum influenza vaccine based upon the internal influenza nucleoprotein (NP) as a target for immune response.

DETAILED DESCRIPTION:
The present study is being conducted in order to generate epidemiological data in support of Osivax's clinical development of a broad spectrum influenza vaccine based upon the internal influenza nucleoprotein (NP) as a target for immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Healthy male or female subjects, as determined by medical history and medical examination (as needed).
3. Between the ages of 18 and 55 years, inclusive.
4. Subject who has fully been vaccinated with licensed severe Acute Respiratory Syndrome SARS-CoV-2 (COVID-19) vaccine(s) according to national recommendations for the corresponding population group.
5. Reliable and willing to make themselves available for the duration of the study, and willing and able to follow study procedures.
6. Ability and technical possibility for completing an electronic Diary (eDiary) and electronic Flu-PRO® questionnaire (ePRO).

Exclusion Criteria:

1. Previous influenza vaccination within 6 months before the day of enrollment or planned to receive during the study duration.
2. Any known or suspected immunodeficient conditions.
3. Current history of significant uncontrolled medical illness such as diabetes, hypertension, heart, renal or hepatic diseases, as judged by the Investigator.
4. Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) to the subject's knowledge.
5. Administration of any investigational or non-registered drug or vaccine within 3 months prior to enrollment, or planned administration of any such product during the whole study period.
6. History of receiving blood, blood components or immunoglobulins within 3 months prior to the day of enrollment, or planned to receive such product during the whole study period.
7. Behavioral or cognitive impairment, or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the study.
8. Past (stopped less than 6 months before enrolment) or current history of alcohol or drug abuse, or current smoking habit above 10 cigarettes per day, or current vaping.
9. Treatment that can affect immune response such as systemic or high dose inhaled corticosteroids (>800μg/day beclomethasone or equivalent; occasional inhaled corticosteroids for asthma therapy are allowed), radiation treatment, cytotoxic drugs, or current or recent (within 30 days before study entry) chronic or prolonged (>10 days) use of systemic non-steroidal antiinflammatory drugs, interferon, immunomodulators, allergy shots, as judged by the Investigator.
10. Individuals with history of any illness that, in the opinion of the Investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects, men and women aged 18 to 55 years.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Proportion of overall subjects reporting Influenza-Like-Illness cases as per Flu-PRO® questionnaire. | Through study completion, an average of 8 months.
Proportion of subjects reporting Influenza-Like-Illness cases as per Flu-PRO® questionnaire with laboratory-confirmed influenza. | Through study completion, an average of 8 months.
Proportion of subjects reporting Influenza-Like-Illness cases as per Flu-PRO® questionnaire with non-laboratory-confirmed influenza. | Through study completion, an average of 8 months.
Severity scores of overall Influenza-Like-Illness cases as per Flu-PRO® questionnaire. | Through study completion, an average of 8 months.
Severity scores of Influenza-Like-Illness cases as per Flu-PRO® questionnaire with laboratory-confirmed influenza. | Through study completion, an average of 8 months.
Severity scores of Influenza-Like-Illness cases as per Flu-PRO® questionnaire with non-laboratory-confirmed influenza. | Through study completion, an average of 8 months.
Duration of overall Influenza-Like-Illness cases as per Flu-PRO® questionnaire. | Through study completion, an average of 8 months.
Duration of Influenza-Like-Illness cases as per Flu-PRO® questionnaire with laboratory-confirmed influenza. | Through study completion, an average of 8 months.
Duration of Influenza-Like-Illness cases as per Flu-PRO® questionnaire with non-laboratory-confirmed influenza. | Through study completion, an average of 8 months.
Anti-NP immunoglobulin G (IgG) titers by ELISA at each time point. | Through study completion, an average of 8 months.
Symptomatic and asymptomatic flu cases based on the abovementioned variables/parameters. | Through study completion, an average of 8 months.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Leroux-Roels, MD, PhD, Principal Investigator — Centre for Vaccinology (CEVAC), Ghent University Hospital
Locations (1):
- Centre for Vaccinology (CEVAC), Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No